CLINICAL TRIAL: NCT00282438
Title: Hematopoietic Stem Cell Transplant in Patients With Refractory Sarcoidosis: A Phase I/II Trial
Brief Title: Hematopoietic Stem Cell Support in Patients With Refractory Sarcoidosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No plan to continue enrollment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU FDA SARC.2003
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous hematopoietic stem cell transplantation (Experimental): Autologous stem cells will be injected after conditioning
  Interventions: Biological: Autologous hematopoietic stem cell transplantation
- Allogeneic stem cell transplantation (Experimental): Allogeneic stem cells will be injected after conditioning
  Interventions: Biological: Allogeneic stem cell transplantation

INTERVENTIONS:
Biological: Autologous hematopoietic stem cell transplantation — Autologous hematopoietic stem cells will be injected after conditioning
  Other Names: Autologous stem cell injection
  Arms: Autologous hematopoietic stem cell transplantation
Biological: Allogeneic stem cell transplantation — Allogeneic stem cells will be injected after conditioning
  Arms: Allogeneic stem cell transplantation

SUMMARY:
Sarcoidosis is a disease believed to be due to immune cells, cells which normally protect the body, but are now attacking lungs, heart, nerves, or other organs or systems within the body. As a result, the affected organs or systems fail to work properly causing difficulty breathing; heart failure; inability of the nerves to respond properly causing numbing, tingling, pain, and progressive muscle weakness; or other symptoms depending on the organ or body system involved. The likelihood of progression of this disease is high. This study is designed to examine whether treating patients with high dose cyclophosphamide (a drug which reduces the function of the immune system) and ATG (a protein that kills the immune cells that are thought to be causing this disease), followed by return of the previously collected blood stem cells will stop the progression of sarcoidosis. Stem cells are undeveloped cells that have the capacity to grow into mature blood cells, which normally circulate in the blood stream. The purpose of the high dose cyclophosphamide and ATG is to destroy the cells in the immune system. The purpose of the stem cell infusion is to evaluate whether this treatment will produce a normal immune system that will no longer attack the body.

DETAILED DESCRIPTION:
Method of Harvesting Stem Cells

Based on the experience of the pilot studies, the current protocol will mobilize stem cells with granulocyte-colony stimulating factor (G-CSF) and collect stem cells by apheresis, with subsequent bone marrow harvest performed only if needed to supplement the peripheral blood stem cells (PBSC). Based on experience of autoimmune flares in patients receiving G-CSF alone for mobilization, patients will be mobilized with cyclophosphamide 2.0 g/m2 and G-CSF 10 mcg/kg.

Cyclophosphamide

Cyclophosphamide (CY) is an active agent in patients with a wide variety of malignancies. It is used frequently in the therapy of lymphoid malignancies and has potent immunosuppressive activity. It is frequently used as a cytotoxic and immunosuppressive agent in patients undergoing marrow transplants and as a treatment for patients with autoimmune diseases. It is an alkylating agent that requires hepatic metabolism to the active metabolites, phosphoramide mustard and acrolein. These active metabolites react with nucleophilic groups. It is available as an oral or intravenous preparation. Bioavailability is 90% when given orally. The half-life of the parent compound is 5.3 hours in adults, and the half-life of the major metabolite phosphoramide mustard is 8.5 hours. Liver or renal dysfunction will lead to prolonged serum half-life. CY is administered intravenously at a dosage of 60 mg/kg on each of 2 successive days (use adjusted ideal body weight if patient's actual body weight is greater than 100% ideal body weight). The major dose limiting side effect at high doses is cardiac necrosis. Hemorrhagic cystitis can occur and is mediated by the acrolein metabolite. This can be prevented by co-administration of MESNA or bladder irrigation. Other notable side effects include nausea, vomiting, alopecia, myelosuppression and SIADH. Refer to institutional manuals for more information about administration, toxicity and complications.

Rabbit-Derived Anti-Thymocyte Globulin (ATG)

Rabbit-derived anti-human thymocyte globulin (ATG) is a gamma globulin preparation obtained from hyperimmune serum of rabbits immunized with human thymocytes. ATG has been used predominately in solid organ transplant immunosuppressive regimens. ATG is a predominantly lymphocyte-specific immunosuppressive agent. It contains antibodies specific to the antigens commonly found on the surface of T cells. After binding to these surface molecules, ATG promotes the depletion of T cells from the circulation through mechanisms, which include opsonization and complement-assisted, antibody-dependent, cell-mediated cytotoxicity. The plasma half-life ranges from 1.5 12 days. ATG is administered intravenously at a dose of 0.5-mg/kg recipient body weight on day -6 and at a dose of 1.0 mg/kg recipient body weight on days -5 to -1. Unlike equine ATG, rabbit ATG does not require a pre-infusion skin test to check for hypersensitivity. Methylprednisolone 250mg (dose adjusted based on patient's condition) will be given before every dose of ATG. Additional medications such as diphenhydramine may be given at the discretion of the attending physician. Although rare, the major toxicity is anaphylaxis; chills, fever, pruritus or serum sickness may occur.

Fludarabine

Fludarabine phosphate is rapidly dephosphorylated to 2-fluoro-ara-A and then phosphorylated intracellularly by deoxycytidine kinase to the active triphosphate, 2-fluoro-ara-ATP. This metabolite appears to act by inhibiting DNA polymerase alpha, ribonucleotide reductase and DNA primase, thus inhibiting DNA synthesis. The mechanism of action of this antimetabolite is not completely characterized and may be multi-faceted.

Phase I studies in humans have demonstrated that fludarabine phosphate is rapidly converted to the active metabolite, 2-fluoro-ara-A, within minutes after intravenous infusion. Consequently, clinical pharmacology studies have focused on 2-fluoro-ara-A pharmacokinetics. After the five daily doses of 25 mg 2-fluoro-ara-AMP/m2 to cancer patients infused over 30 minutes, 2-fluoro-ara-A concentrations show a moderate accumulation. During a 5-day treatment schedule, 2-fluoro-ara-A plasma trough levels increased by a factor of about 2. The terminal half-life of 2-fluoro-ara-A was estimated as approximately 20 hours. In vitro, plasma protein binding of fludarabine ranged between 19% and 29%.

CAMPATH

Campath-1H is a humanized fusion protein that is directed to CD52 antigen that is expressed on all lymphocytes, monocytes and macrophages. It has very potent immunosuppressive property and is effective for prevention of graft-versus-host disease. 30 mg/day of CAMPATH will be given intravenously over 2 hours on days -4, -3 and -2. The most commonly reported adverse reactions are infusion reactions fever, chills, hypotension, urticaria, nausea, rash, tachycardia, dyspnea), cytopenias (neutropenia, lymphopenia, thrombocytopenia, anemia), and infections (CMV viremia, CMV infection, other infections). In clinical trials, the frequency of infusion reactions was highest in the first week of treatment. Other commonly reported adverse reactions include vomiting, abdominal pain, insomnia and anxiety. The most commonly reported serious adverse reactions are cytopenias, infusion reactions, and immunosuppression/infections. About 30 minutes before the patient gets Campath, he/she will be given other medications (such as acetaminophen or diphenhydramine, given orally, not IV) to help reduce side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18years and ≤ 60 years at the time of pretransplant evaluation.
2. Definitive diagnosis of sarcoidosis in pathologic specimen.
3. Patients who failed to respond to conventional treatment of at least 3 months duration with corticosteroids (equivalent dosage of prednisone 1.0mg/kg/day to start). Patients must also have failed two or more of the followings: TNF inhibitors (etanercept, infliximab), methotrexate, azathioprine, 6-MP, cyclosporin, tacrolimus, mycophenolate mofetil, gold, dapsone, colchicine, chloroquine/hydroxychloroquine or any other immunosuppressive or modulating drugs.
4. Failure of therapy defined by (not caused by unrelated conditions) any one of following:

   * Progressive pulmonary disease (stage II or III) defined by decline in pulmonary function (DLCo, VC or FEV1) of 15% or more over 12 months.
   * Progressive CNS disease (worsening symptoms such as paraparesis or medically refractory seizure).
   * Persistent peripheral neuropathy (one of following):

     1. Persistent muscle weakness Grade 3/5 or worse (MRC) in at least one movement (e.g. ankle dorsiflexion) in two limbs.
     2. Persistent cranial nerve involvement such as persistent facial diplegia.
     3. Persistent incapacitating sensory loss (e.g. gait ataxia, falls > 1/month).
   * Progressive loss of vision.
   * Persistent hypercalcemia.
5. Cardiac sarcoidosis that is proven by cardiac biopsy or cardiac MRI.

Exclusion Criteria:

1. Alternative diagnosis.
2. Noncompliance to medical care.
3. > 10 pack-year history of cigarette smoking if lung disease is the major problem.
4. Poor performance (PS) status (ECOG >2) at the time of entry, unless decline of PS is due to the disease itself.
5. Significant end organ damage such as:

   1. Overt congestive heart failure (NYHA Class III or IV).
   2. Active ischemic heart disease, s/p myocardial infarction within 6 months, s/p unstable angina within 3 months, s/p CVA within 6 months, s/p hospitalization for CHF within 3 months.
   3. Untreated life-threatening arrhythmia.
   4. Pulmonary hypertension > 40 mmHg.
   5. End-stage lung disease (TLC < 55%, FVC < 55%, or DLCO < 40% of predicted value).
   6. Serum creatinine > 2.5 or creatinine clearance < 30 ml/min.
   7. Liver cirrhosis, transaminases > 3x normal or bilirubin > 2.0 unless due to Gilbert's disease.
6. HIV positive.
7. Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment.
8. Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis.
9. Positive pregnancy test, inability or unable to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
10. Significant psychological issues, social issues, psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
11. Inability to give informed consent.
12. Major hematological abnormalities such as platelet count less than 100,000/ul, ANC less than 1000/ul.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2003-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autologous Hematopoietic Stem Cell Transplantation | Allogeneic Stem Cell Transplantation
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Hematopoietic Stem Cell Transplantation | Allogeneic Stem Cell Transplantation | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (NA) — Only one participant was analyzed and then the standard deviation could only be provided for the total column. | 49 (NA) — Only one participant was analyzed and then the standard deviation could only be provided for the total column | 51.5 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Presence of Toxicity
Description: Daily assessment will be made with regards to toxicity by one of the protocol investigators.National Cancer Institute Common Toxicity Criteria will be used to grade all non-hematologic toxicities. Toxicity grades as follows: 1 = Mild; 2 = Moderate; 3 = Severe and undesirable; 4 = life threatening or disabling ; 5 = Death
Time Frame: For length of hospital stay (until discharge).
Measure: Number; unit: participants
Arm/Group | Autologous Hematopoietic Stem Cell Transplantation | Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 1 | 1
participants | 1 | 1

2. Primary Outcome: Survival
Description: Patient has not died.
Time Frame: Participants are to be followed at 6 months and then yearly until 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous Hematopoietic Stem Cell Transplantation | Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

3. Primary Outcome: Time to Disease Progression
Description: Worsening symptoms, pulmonary function studies, cardiac function and arrhythmia including EKG assessments, and neurological symptoms.
Time Frame: Participants are to be followed at 6 months and then yearly until 5 years
Measure: Number; unit: months
Arm/Group | Autologous Hematopoietic Stem Cell Transplantation | Allogeneic Stem Cell Transplantation
Number analyzed (Participants) | 1 | 1
months | 4 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of first transplant 4/25/2012 until patient death 6/27/2015. Study closure effective 8/17/2015.
Arm/Group | Autologous Hematopoietic Stem Cell Transplantation | Allogeneic Stem Cell Transplantation
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Hematopoietic Stem Cell Transplantation (N=1) | Allogeneic Stem Cell Transplantation (N=1)
Death (Infections and infestations) | 0 (0) | 1 (1) — 70 days after the transplant developed staphylococcus aureus sepsis, complicated by ARDS and respiratory failure
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — 70 days after the transplant developed staphylococcus aureus sepsis, complicated by ARDS and respiratory failure

LIMITATIONS AND CAVEATS:
Two patients had been enrolled on trial. One underwent autologous HSCT and relapsed early after the transplant. The second participant underwent allogeneic HSCT and died 70 days after the transplant and the study has been terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No